CLINICAL TRIAL: NCT06995222
Title: The Role of Renal Resistive Index (RI) in Predicting Acute Kidney Injury Progression and Need for Renal Replacement Therapy in Patients Followed in the Intensive Care Clinic
Brief Title: The Role of Renal Resistive Index (RI) in Predicting Acute Kidney Injury Progression in Intensive Care Clinic
Status: Recruiting | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mete Erdemir, principal investigator, Gulhane Training and Research Hospital
Other Study IDs: 2025-07
Record Dates: First submitted 2025-04-04; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Akut Kidney Injury; Renal Replacement Therapy for Acute Kidney Injury in ICU
Keywords: akut kidney injury; renal resistive index; renal replacement therapy; intensive care
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: renal resistive index with Doppler ultrasound — Renal resistive index uses doppler ultrasonography which assesses blood flow velocity in the renal arteries. The Renal Resistive Index (RI) is calculated by substracting diastolic velocity from systolic velocity then dividing result by systolic velocity
  Where:
  Systolic velocity is the peak velocity of the blood flow during the systolic phase of the cardiac cycle.
  Diastolic velocity is the velocity of blood flow during the diastolic phase.

SUMMARY:
Acute kidney injury(AKI) is defined in the KDIGO guidelines as a ≥0.3 mg/dL (≥26.5 micromol/L) increase in serum creatinine in the previous 48 hours or a ≥1.5-fold increase in serum creatinine from baseline, known or presumed to have occurred in the previous seven days, or a urine volume <0.5 mL/kg/hour for six hours.

Given the high morbidity and mortality associated with AKI, many investigators are studying several novel biomarkers to detect AKI progression earlier, identify etiologies and predict outcomes. However, the utilisation of these novel biomarkers may be constrained by reimbursement considerations.

The renal resistive index (RRI) is a well-established metric for evaluating renal perfusion; however, its application in the context of AKI has been a subject of recent debate. While RRI has been utilised to demonstrate perfusion in acute and chronic renal diseases, particularly in conjunction with ultrasonography, its efficacy remains a subject of scientific discourse. In addition, Boddi reported that RRI is a strong indicator of mortality and a diagnostic marker, especially in patients with persistent AKI.

The present study aims to evaluate the appropriateness of using the RRI, a non-invasive procedure, to determine the progression of AKI stages and the need for renal replacement therapy in patients hospitalised in intensive care units.

DETAILED DESCRIPTION:
Acute kidney injury(AKI) KDIGO guidelines for AKI include an increase in serum creatinine of ≥0.3 mg/dL (≥26.5 micromol/L) in the last 48 hours or an increase in serum creatinine of ≥1 mg/dL (≥26.5 micromol/L) from baseline, known or presumed to have occurred in the previous seven days, 5-fold increase or urine volume <0.5 mL/kg/hour for six hours.

The incidence of in-hospital AKI varies between 7. 0-18.3% in hospitalized patients in general and up to 20-50% in critically ill patient populations . In addition to causing a high mortality and morbidity, especially in critically ill patients, AKI prolongs the duration of hospitalization in the intensive care unit.

Due to the high morbidity and mortality associated with AKI, many researchers have been studying several novel biomarkers for earlier detection of AKI progression, identification of etiologies and prediction of outcomes. However, the use of these new biomarkers may be limited by reimbursement issues.

Although renal resistive index(RRI) shows intraparenchymal perfusion of the kidney, RRI is used to show perfusion in acute and chronic diseases of the renal parenchyma, especially as a result of the widespread use of ultrasonography(USG) in recent times. In addition, Boddi reported that RRI is a strong indicator of mortality and a diagnostic marker, especially in patients with persistent AKI. Many studies have shown that RRI is a promising marker for early detection of renal injury. Patients who develop AKI often require renal replacement therapy (RRT), but there is generally no consensus on the optimal timing of the initiation of RRT. RRT is an invasive procedure. The desired outcome in patients with AKI is normalization of renal function without invasive intervention. However, a more conservative approach to initiating RRT in the course of AKI may expose the patient to adverse outcomes. Therefore, designing a marker that predicts the likelihood of a more severe AKI progression would help us to better make decisions regarding the optimal timing of RRT initiation.

In this study, we aimed to evaluate the appropriateness of using the RRI, a noninvasive procedure, to detect progression in AKI stages and the need for RRT in intensive care unit patients.

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years of age
2. Having KDIGO stage 1 or stage 2 acute kidney injury within the first 24 hours of admission

Exclusion Criteria:

* 1. Patients who did not provide a consent form for participation in the study 2. Patients under 18 years of age 3. Pregnant women 4. Patients with postrenal acute kidney injury 5. Patients 24 hours after the diagnosis of acute kidney injury 6. Patients with acute kidney injury in the recovery period 7. Patients who were evaluated as KDIGO ABH stage 3 during hospitalization 8. Patients with a known history of renal artery stenosis 9. Patients with a diagnosis of cardiac arrhythmia 10. Patients with a diagnosis of chronic kidney disease and a glomerular filtration rate below 30 ml/min/1.73m2 11. Patients with intra-abdominal pressure above 20 mmHg 12. Patients with a hospitalization period of less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients over 18 years of age who met KDIGO ABH stage 1 or stage 2 criteria and were hemodynamically stable in the first 24 hours of admission to the Internal Medicine Intensive Care Unit of Gülhane Training and Research Hospital, University of Health Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Akut kidney injury progression | 14 days
  Patients admitted to our intensive care clinic with a diagnosis of AKI stage 1-2(according to KDIGO staging) will have RI measurement with Doppler Ulsanography within the first 24 hours of admission. Patients will be followed up daily from the time of measurement until the end of the study period and their progression to AKI stage 3(according to KDIGO staging) will be recorded. Patients will be monitored throughout the study. A comparison will be made between the groups that developed AKI stage 3(according to KDIGO staging) and those that did not develop AKI stage 3 during the study.

SECONDARY OUTCOMES:
14th day mortality rate | 14 days
  The mortality status of patients on the 14th day after ICU admission will be recorded. The relationship between RI value and 14-day mortality will be evaluated.
28th day mortality rate | 28 days
  The mortality status of patients on the 28th day after ICU admission will be recorded. The relationship between RI value and 28-day mortality will be evaluated.
Length of stay in the intensive care unit | 18 months
  The duration of stay in the ICU will be recorded for each patient. The association between RI value and length of ICU stay will be assessed.
Need for renal replacement therapy (RRT) | 14 days
  The requirement for RRT during ICU stay will be recorded according to KDIGO criteria. Patients who require RRT will be compared with those who do not, in terms of RI level.

CONTACTS AND LOCATIONS:
Overall Officials: Gürhan T associate professor doctor, Study Director — Gulhane Education and Research Hospital Ankara Türkiye
Locations (1):
- Gulhane Education and Research Hospital Ankara Türkiye, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
research results will be published and the data used in the publication will be available for sharing upon request
Supporting Information: Study Protocol
Time Frame: January 01, 2025 - July 01, 2026
Access Criteria: During the publication phase, it will be shared with the relevant broadcasting organization via the official e-mail address, and patient identification information will not be specified.

REFERENCES:
- [Background] Gibney N, Hoste E, Burdmann EA, Bunchman T, Kher V, Viswanathan R, Mehta RL, Ronco C. Timing of initiation and discontinuation of renal replacement therapy in AKI: unanswered key questions. Clin J Am Soc Nephrol. 2008 May;3(3):876-80. doi: 10.2215/CJN.04871107. Epub 2008 Mar 5. PMID 18322044